CLINICAL TRIAL: NCT01955044
Title: Early DHA Supplementation in Extremely Low Birth Weight Infants
Brief Title: PUFA Supplementation in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Northwestern University Feinberg School of Medicine (Other); Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Brandy Frost, Attending Neonatologist, Clinician Educator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EH13-334
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Premature, Extremely Low Birth Weight Infants; Polyunsaturated Fatty Acid Levels
Keywords: neonatal prematurity; infant, extremely low birth weight; fatty acids, polyunsaturated
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "high" dose LCPUFA (Experimental): the "high" dose LCPUFA supplement is a drop that will be administered to ELBW infants.
  Interventions: Dietary Supplement: LCPUFA supplement
- "low" dose LCPUFA (Experimental): the "low" dose LCPUFA supplement is a drop that will be administered to ELBW infants.
  Interventions: Dietary Supplement: LCPUFA supplement
- placebo (Placebo Comparator): the "placebo" is a drop that will be administered to ELBW infants.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: LCPUFA supplement
  Other Names: PUFA supplement
  Arms: "high" dose LCPUFA; "low" dose LCPUFA
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if buccal administration of a concentrated formulation of long-chain polyunsaturated fatty acids (LCPUFA) can help to maintain docosahexaenoic acid (DHA) levels in extremely low birth weight (ELBW) infants.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, placebo controlled, double blind trial.

Two doses of PUFA will be compared to placebo- a "high" dose and a "low" dose.

ELBW infants will be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* a) Premature infant born at gestational age less than 34 weeks
* b) Birth weight less than 1000 grams
* c) Legally authorized representative is able to provide written informed consent within the first 72 hours of life, prior to the performance of an protocol-specified evaluations or procedures

Exclusion Criteria:

* a) infants with known metabolic disorder
* b) infants with known congenital gastrointestinal anomaly
* c) infants who are deemed to be inappropriate for enrollment per attending neonatologist

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Caplan, MD, Principal Investigator — Endeavor Health
Locations (3):
- United States (3):
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Prentice Women's Hospital, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

REFERENCES:
- [Derived] Robinson DT, Caplan M, Carlson SE, Yoder R, Murthy K, Frost B. Early docosahexaenoic and arachidonic acid supplementation in extremely-low-birth-weight infants. Pediatr Res. 2016 Oct;80(4):505-10. doi: 10.1038/pr.2016.118. Epub 2016 Jun 3. PMID 27356083

RESULTS

PARTICIPANT FLOW:
Groups:
- "High" Dose LCPUFA: the "high" dose LCPUFA supplement is a drop that will be administered to ELBW infants.
  LCPUFA supplement
- "Low" Dose LCPUFA: the "low" dose LCPUFA supplement is a drop that will be administered to ELBW infants.
  LCPUFA supplement
- Placebo: the "placebo" is a drop that will be administered to ELBW infants.
  placebo
Period: Overall Study
Arm/Group | "High" Dose LCPUFA | "Low" Dose LCPUFA | Placebo
Started | 10 | 10 | 10
Completed | 9 | 9 | 10
Not Completed | 1 | 1 | 0
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "High" Dose LCPUFA | "Low" Dose LCPUFA | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 10 | 30
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 11
  Male | 8 | 5 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Long-chain Polyunsaturated Fatty Acid (LCPUFA) Levels
Description: LCPUFA levels will be measured at 2 weeks of life in extremely low birth weight (ELBW) infants
Time Frame: 2 weeks of life
Population: 2 subjects died prior to having 2 week levels drawn, from causes unrelated to study.
Measure: Median (Inter-Quartile Range); unit: weight % (g/100g)
Arm/Group | "High" Dose LCPUFA | "Low" Dose LCPUFA | Placebo
Number analyzed (Participants) | 9 | 9 | 10
weight % (g/100g)
  2 week DHA levels | 4.45 [4.36 to 5.16] | 4.02 [3.96 to 4.77] | 5.27 [4.75 to 5.63]
  2 week ARA (arachidonic acid) levels | 20.3 [18.91 to 21.34] | 19.3 [17.64 to 22.54] | 21.58 [20.2 to 23.04]

2. Secondary Outcome: LCPUFA Levels
Description: LCPUFA levels will be measured at 8 weeks of life.
Time Frame: 8 weeks of life
Population: 2 subjects died prior to having 8 week levels drawn, from causes unrelated to study.
Measure: Median (Inter-Quartile Range); unit: wt% (g/100g)
Arm/Group | "High" Dose LCPUFA | "Low" Dose LCPUFA | Placebo
Number analyzed (Participants) | 9 | 9 | 10
wt% (g/100g)
  8 week DHA levels | 5.52 [4.45 to 7.08] | 5.58 [5.49 to 6.96] | 6.75 [5.22 to 7.4]
  8 week ARA levels | 19.79 [17.77 to 22.99] | 19.9 [18.3 to 21.06] | 22.21 [19.05 to 23.11]
Statistical Analysis 1: Comparison: "High" Dose LCPUFA vs "Low" Dose LCPUFA vs Placebo; DHA levels; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.23

ADVERSE EVENTS:
Arm/Group | "High" Dose LCPUFA | "Low" Dose LCPUFA | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "High" Dose LCPUFA (N=10) | "Low" Dose LCPUFA (N=10) | Placebo (N=10)
death (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Baby died from NEC, deemed unrelated to study substance
death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — severe respiratory failure
spontaneous bowel perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No